CLINICAL TRIAL: NCT05848505
Title: Effect of Preoperative Intranasal Dexmedetomidine on Fentanyl Requirements in Children Undergoing Tonsillectomy
Brief Title: Opioid-sparing Effect of Intranasal Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre-Yves P Lequeux (Other)
Responsible Party: Sponsor-Investigator, Pierre-Yves P Lequeux, Consultant aneshesiologist, Sheikh Khalifa Medical City
Organization: Sheikh Khalifa Medical City (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-08.02.2022 [RS-741]
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Tonsillar Hypertrophy
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): Intranasal dexmedetomidine 2 mcg/kg administered before surgery
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Intranasal saline 0.02 mL/kg administered before surgery
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal administration Dosage 2 mcg/kg

SUMMARY:
Background: Management of postoperative pain in paediatric patients undergoing tonsillectomy remains a challenge that faces anesthesiologists in their daily practice. High dose of opioids are usually necessary and are responsible for side effects like nausea, vomiting, constipation, delayed hospital discharge and more importantly respiratory depression and sleep apnea. Dexmedetomidine is a selective alpha two agonist that has an analgesic and anxiolytic effect with minimal effects on respiratory drive.

Goal of the study: The aim of this study is to assess the opioid sparing effect of preoperative intranasal dexmedetomidine as part of multimodal analgesia in the paediatric population undergoing tonsillectomy.

Methods: This will be a prospective, randomised, controlled, double blinded clinical trial with 50 participants who will be randomised between two groups: dexmedetomidine group and control group. The dexmedetomidine group will receive intranasal dexmedetomidine in the preoperative holding area while the other group will receive the placebo.

The primary endpoint will be the total fentanyl consumption in the perioperative period. Additionally, we will look at postoperative pain scores at 10, 30 and 60 minutes after recovery as well as the time to first opioid rescue analgesic and agitation scores as secondary endpoints. Blood pressure and hart rate will also be recorded throughout the study period.

DETAILED DESCRIPTION:
Tonsillectomy surgery is both common and painful in paediatric patients, usually requiring high doses of opioids, which are associated with many adverse effects. Dexmedetomidine is a sedative intravenous drug with analgesic and opioid-sparing effects but with side effects including (usually minor) bradycardia and hypotension which might delay hospital discharge. Intranasal dexmedetomidine, although off-label, has been extensively studied for its sedative effect as well as its safety profile and is associated with much less side effects (bradycardia and hypotension). It has however not being studied for its analgesic effects in children. The hypothesis is that preoperative intranasal dexmedetomidine will decrease total perioperative fentanyl consumption in children undergoing tonsillectomy.

Fifty ASA 1 or 2 patients aged from 3 yo to 6 yo scheduled for tonsillectomy (+/- adenoidectomy +/- myringotomy) will be included in this prospective, randomised, controlled, double blind trial and then randomised in two groups: dexmedetomidine group (DG) and control group(CG).

Exclusion criteria are: allergy to dexmedetomidine, paracetamol, ondansetron or dexamethasone, hepatic dysfunction, raised intracranial pressure or altered GCS or neuromuscular disease in addition to abnormal neurological development.

Upon arrival in the operating theater holding area, the patients will receive either 2mcg/kg of dexmedetomidine (DG) or the equivalent volume of normal saline (CG), both administered intranasally with a mucosal atomizer device attached to the syringe and equally distributed in both nostrils. Although intranasal dexmedetomidine is off-label, it is routinely administered as a premedication including in our institution. The syringes of dexmedetomidine and normal saline will be prepared by a nurse and both the patients and the anaesthetists will be blinded of the content of the syringes. The patients will then be moved to the operating room and a proper monitoring will be applied (ECG, pulse oximeter, non-invasive blood pressure and capnograph). Anaesthesia will be induced with inhalation of Sevoflurane without nitrous oxide and fentanyl 1 mcg/kg as well as a neuromuscular blocking agent (at the discretion of the anaesthetist) will all be administered as soon as an intravenous cannula is inserted. The trachea will then be intubated before the start of surgery. During the surgery, the anaesthetist in charge will give boluses of 1 mcg/kg of fentanyl when deemed necessary (tachycardia, hypertension, movements of the patient). All the patients will receive the usual analgesia regimen of SKMC consisting of paracetamol (15 mg/kg), dexamethasone (0.15 mg/kg) and ondansetron (0.1 mg/kg) before extubation.

In the Post-Anaesthesia Care Unit (PACU), the patients will be administered 0.5 mcg/kg of fentanyl q10min if their pain score (measured by the FLACC scale) is > 2/10 and repeated until the score is < 3. The PACU nurses will be blinded to which group the patients belong.

The patrients will be randomised in two arms, randomised 1:1, the dexmedetomidine arm (DG) and the control arm (CG). The patients of the DG will receive 2 mcg/kg of dexmedetomidine while the patients of the CG will receive normal saline instead, both will be administered intranasally with a mucosal atomiser device and equally distributed in each nostril. The sample size calculation was made according to the available literature on the opioid-sparing effect of intranasal dexmedetomidine with a type I error rate (alpha) of 5% and a type II error rate (power) of 80%. The result is 25 patients in each arm.

Demographic data will be compared between CG and DG with a Student's t-test or a Chi-square test when appropriate. The total fentanyl consumption as well as the pain and agitation scores of the DG and the CG will be compared using a Student's t-test for mean comparison. A p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective tonsillectomy

Exclusion Criteria:

* documented allergy to dexmedetomidine, paracetamol, ondansetron or dexamethasone
* hepatic dysfunction
* raised intracranial pressure or altered GCS
* neuromuscular disease.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Perioperative fentanyl consumption | From induction of anesthesia to discharge of post-anesthesia care unit (expected less than 4 hours)
  Cumulative perioperative (intraoperative and postoperative) fentanyl consumption

SECONDARY OUTCOMES:
Postoperative pain | From admission to discharge of post-anesthesia care unit (expected less than 3 hours)
  Pain score at 10, 30 and 60 minutes after arrival in the post-anesthesia care unit using the FLACC Scale
Postoperative sedation | From admission to discharge of post-anesthesia care unit (expected less than 3 hours)
  Sedation-agitation score 30 minutes after the arrival in the post-anesthesia care unit using the Riker scale
Post-anesthesia care unit length of stay | From admission to discharge of post-anesthesia care unit (expected less than 3 hours)
  Post-anesthesia care unit length of stay
Bradycardia | From induction of anesthesia to discharge of post-anesthesia care unit (expected less than 4 hours)
  Incidence of intraoperative and postoperative bradycardia defined as heart rate below 70 bpm
Hypotension | From induction of anesthesia to discharge of post-anesthesia care unit (expected less than 4 hours)
  Incidence of intraoperative and postoperative hypotension defined as systolic blood pressure below 70 mmHg + [age x 2] or below 90 mmHg for patients older than 10 year old

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Khalifa Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided